





Institutional Review Board Faculty of Medicine Minia University

Approval No. 99-2021

27<sup>th</sup> September 2021 Hemmat Amer Mohamed Department of Anesthesia & Intensive Care Faculty of Medicine Minia University Egypt

MSC Thesis Title: validity of ultrasonography in predicting difficult laryngoscopy and confirming endotracheal intubation in obese emergency surgical patients.

## Dear | Hemmat Amer Mohamed,

You are kindly informed that this letter has been issued to officially notify you that our Institutional Review Board "IRB", Faculty of Medicine, Minia University, has reviewed & approved your submitted research study documents.

Please note that, as being the principle investigator, you have to:

- 1. Implement this study as of the date of issue of this approval letter.
- 2. Submit any amendments to the approved protocol.
- 3. Submit follow up reports every 6 months.
- 4. Submit an end of study report.

Sincerely,

Associate Prof. Manal Ismail Abd-Elghany, MD (Egypt), PhD (UK)

Associate Professor of Pathology

Manal 9 Abd Elghany

Chairman of Institutional Review Board "IRB"

Faculty of Medicine, Minia University, Egypt

Cell Phone No: +201005765568

Email: manalismail2000@yahoo.co.uk /manal.abdelghany@mu.edu.eg

The Instructional Review Board of Faculty of Medicine, Minia University is constituted and operating according to Declaration of Helsinki, CIOMS, ICH-GCP guidelines, Egyptian law No.214 (2020), and applicable local & institutional guidelines which govern EC operations

Page 1 of 1